CLINICAL TRIAL: NCT00916903
Title: Genetic Disease Gene Identification
Status: Terminated | Type: Observational
Why Stopped: Lack of funding.
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: IRBPHS#4280F
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2024-01-02 (Actual); Status verified 2016-04

CONDITIONS: Congenital Vertical Talus; Familial Encephalopathy With Neuroserpin Inclusion Bodies; Idiopathic Generalised Epilepsy; Familial Dementia; X-linked Mental Retardation
Keywords: Talus; Neuroserpin; mental retardation; epilepsy; FENIB; XLMR
MeSH Terms: conditions — Flatfoot; Familial encephalopathy with neuroserpin inclusion bodies; Epilepsy, Idiopathic Generalized; Dementia; X-Linked Intellectual Disability; Intellectual Disability; Epilepsy

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA will be isolated from peripheral blood or cheek scraoes.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients with genetic condition being studied.
- 2: Matched controls

SUMMARY:
This is a a study to identify inherited disease genes. The study will use molecular techniques to map genetic diseases using techniques such as Affymetrix SNP chips. The powerful combination of the information generated by the Human Genome Project and technical advances such as microarrays enables attempts to identify genes responsible for inherited disorders more possible than ever before. Starting with even modest pedigrees of only a few individuals, or even single individuals, it is possible to identify the gene(s) involved. It is proposed to collect up to 20 ml of peripheral blood and/or buccal cell samples from subjects and relevant family members. Currently the following disorders are approved for investigation.

The current list of disorders:

Aarskog-Scott syndrome, Café-au-Lait spots, Cerebral cavernous malformation, delXp, del2q, del10p, del11q, del12p, del13q, del14q, del16q, del17q, del18q, del Xp21, Choreoathetosis, Congenital Vertical Talus (CVT), Clubfoot, Tarsal coalition and other congenital limb deformities, Cystic Fibrosis (CF)-like disease, Desbuquois syndrome, Droopy Eyelid syndrome (Ptosis), Fanconi-Bickel syndrome (FBS), FENIB (familial encephalopathy with neuroserpin inclusion bodies), FG syndrome, Idiopathic generalised epilepsy (IGE), Renpenning syndrome, transient neonatal diabetes with 6q UPD, translocation (13;14), translocation (3;8), translocation (2;18), Uncharacterized familial dementia and X-linked mental retardation (XLMR).

DETAILED DESCRIPTION:
It is proposed to identify and recruit individuals and/or families with specified the disorders listed above. 10-20 ml (2-4 teaspoons) of peripheral blood will be collect¬ed from all adult subjects. Smaller volumes of blood would be collected from children based on their age/size. In some cases, as an adequate alternative to collecting peripheral blood, buccal cells will be collected using cheek swabs (Epicentre Biotechnologies). All relevant living members of each pedigree will be asked to partici¬pate, free of charge, on a research basis only. Genomic DNA will be extracted by standard methods and used as template for Polymerase Chain Reac¬tion (PCR) amplification reactions. Individuals will be genotyped at markers and candidate gene sequenced.

Essentially two approaches will be used:

1. Circumstances that may provide knowledge of candidate genes include reviews of the literature, biology of the disease, understanding of biological pathways, chromosomal rearrangements, mutants in model organisms etc. When candidate genes exist, it is proposed to use linked microsatellite and/or single nucleotide polymorphism (SNP) PCR primer pairs on the DNA from families to determine if there is co-segregation of the disease and markers and thus linkage between the disease gene and previously mapped markers.

   If the disease appears to be linked to the candidate gene, PCR primers flanking all coding exons will be used to amplify the exons and intron/exon boundaries followed by sequencing to detect disease-causing mutations. A web site that enables the design of primers to amplify candidate gene exons is available (http://genome.ucsc.edu/cgi-bin/hgGateway ). If a very strong candidate gene exists, candidate gene sequencing will be performed on affected individual samples without first performing a linkage study.
2. When no obvious candidate genes exist, and a family of sufficient size has been collected, it is proposed to use Affymetrix SNP microarrays to perform a human genome-wide search for linkage. We have used this approach successfully before (Shrimpton et al 2004), utilizing the whole genome linkage analysis with the Human Mapping 10K Array (Affymetrix Inc., Santa Clara, CA). The 10K Array permits the simultaneous genotyping of more than 11,200 mapped SNPs spaced throughout the human genome at 210 KB intervals. Affymetrix 100K and 500K arrays are also available. SNP genotype information will be analyzed using Varia (Silicon Genetics) and/or Merlin software. The data will be used to define a critical region. If statistically significant segregation is detected, candidate genes within the critical region will be evaluated and ranked in order of their likelihood of being the disease gene. Candidate genes will then be sequenced as detailed above.

Summary.

1. Identify candidate disease genes from linkage studies, strong circumstantial evidence or clues from the phenotype.
2. Sequence candidate genes to detect disease-causing mutations.
3. Evaluation of detected variation.

ELIGIBILITY:
Inclusion Criteria:

* Patients and their families identified by physicians.

Exclusion Criteria:

* Patients with unrelated disorders.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients and their families identified by physicians.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2005-10; Primary Completion 2015-04 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Identification of gene/mutation responsible for disorder. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Antony E Shrimpton, PhD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

REFERENCES:
- [Background] Shrimpton AE, Levinsohn EM, Yozawitz JM, Packard DS Jr, Cady RB, Middleton FA, Persico AM, Hootnick DR. A HOX gene mutation in a family with isolated congenital vertical talus and Charcot-Marie-Tooth disease. Am J Hum Genet. 2004 Jul;75(1):92-6. doi: 10.1086/422015. Epub 2004 May 14. PMID 15146389
- [Background] Bradshaw CB, Davis RL, Shrimpton AE, Holohan PD, Rea CB, Fieglin D, Kent P, Collins GH. Cognitive deficits associated with a recently reported familial neurodegenerative disease: familial encephalopathy with neuroserpin inclusion bodies. Arch Neurol. 2001 Sep;58(9):1429-34. doi: 10.1001/archneur.58.9.1429. PMID 11559315
- [Result] Hoo JJ, Shrimpton AE. Distal 3p deletion is not necessarily associated with dysmorphic features or psychomotor delay. Am J Med Genet A. 2008 Feb 15;146A(4):538. doi: 10.1002/ajmg.a.32158. No abstract available. PMID 18203205
- [Result] Shrimpton AE, Jensen KA, Hoo JJ. Karyotype-phenotype analysis and molecular delineation of a 3p26 deletion/8q24.3 duplication case with a virtually normal phenotype and mild cognitive deficit. Am J Med Genet A. 2006 Feb 15;140(4):388-91. doi: 10.1002/ajmg.a.31066. No abstract available. PMID 16411192
- [Result] Hoo JJ, Shrimpton AE. Familial hyper- and hypopigmentation with age-related pattern change. Am J Med Genet A. 2005 Jan 15;132A(2):215-8. doi: 10.1002/ajmg.a.30381. No abstract available. PMID 15551335
- [Result] Shrimpton AE, Braddock BR, Thomson LL, Stein CK, Hoo JJ. Molecular delineation of deletions on 2q37.3 in three cases with an Albright hereditary osteodystrophy-like phenotype. Clin Genet. 2004 Dec;66(6):537-44. doi: 10.1111/j.1399-0004.2004.00363.x. PMID 15521982
- [Result] Levinsohn EM, Shrimpton AE, Cady RB, Packard DS, Hootnick DR. Congenital vertical talus in four generations of the same family. Skeletal Radiol. 2004 Nov;33(11):649-54. doi: 10.1007/s00256-004-0851-1. Epub 2004 Sep 11. PMID 15368082
- [Result] Davis RL, Shrimpton AE, Carrell RW, Lomas DA, Gerhard L, Baumann B, Lawrence DA, Yepes M, Kim TS, Ghetti B, Piccardo P, Takao M, Lacbawan F, Muenke M, Sifers RN, Bradshaw CB, Kent PF, Collins GH, Larocca D, Holohan PD. Association between conformational mutations in neuroserpin and onset and severity of dementia. Lancet. 2002 Jun 29;359(9325):2242-7. doi: 10.1016/S0140-6736(02)09293-0. PMID 12103288
- [Result] LaDine BJ, Simmons JA, Shrimpton AE, Hoo JJ. Syndrome of short stature, widow's peak, ptosis, posteriorly angulated ears, and joint problems: exclusion of the Aarskog (FGD1) gene as a candidate gene. Am J Med Genet. 2001 Mar 15;99(3):248-51. doi: 10.1002/1096-8628(2001)9999:99993.0.co;2-t. PMID 11241498
- [Result] Shrimpton AE, Braddock BR, Hoo JJ. Narrowing the map of a gene (MRXS9) for X-linked mental retardation, microcephaly, and variably short stature at Xq12-q21.31. Am J Med Genet. 2000 May 15;92(2):155-6. No abstract available. PMID 10797443
- [Result] Davis RL, Shrimpton AE, Holohan PD, Bradshaw C, Feiglin D, Collins GH, Sonderegger P, Kinter J, Becker LM, Lacbawan F, Krasnewich D, Muenke M, Lawrence DA, Yerby MS, Shaw CM, Gooptu B, Elliott PR, Finch JT, Carrell RW, Lomas DA. Familial dementia caused by polymerization of mutant neuroserpin. Nature. 1999 Sep 23;401(6751):376-9. doi: 10.1038/43894. PMID 10517635
- [Result] Shrimpton AE, Daly KM, Hoo JJ. Mapping of a gene (MRXS9) for X-linked mental retardation, microcephaly, and variably short stature to Xq12-q21.31. Am J Med Genet. 1999 May 28;84(3):293-9. PMID 10331611
- [Result] Davis RL, Holohan PD, Shrimpton AE, Tatum AH, Daucher J, Collins GH, Todd R, Bradshaw C, Kent P, Feiglin D, Rosenbaum A, Yerby MS, Shaw CM, Lacbawan F, Lawrence DA. Familial encephalopathy with neuroserpin inclusion bodies. Am J Pathol. 1999 Dec;155(6):1901-13. doi: 10.1016/S0002-9440(10)65510-1. PMID 10595921